CLINICAL TRIAL: NCT04476589
Title: Prognostication of Recovery in Early Disorders of Consciousness After COVID-19
Acronym: PREDICT-COVID
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian L. Edlow, M.D., Neurocritical Care Faculty, Massachusetts General Hospital
Other Study IDs: 2020P001616
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Covid19; Coma; Consciousness Disorder
MeSH Terms: conditions — COVID-19; Coma; Consciousness Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Disorders of Consciousness: Patients with COVID-19 and disorders of consciousness
  Interventions: Diagnostic Test: Functional MRI

INTERVENTIONS:
Diagnostic Test: Functional MRI — measurement of functional brain networks

SUMMARY:
The primary aim of this research proposal is to use multimodal metrics (e.g., clinical data and advanced neuroimaging) in the early (i.e., acute hospitalization) phase of recovery from COVID-19-related disorders of consciousness to predict outcome at 3, 6, and 12 months post-hospitalization. We aim to construct an algorithm that synthesizes the results of these metrics to help predict recovery.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older,
2. positive diagnosis of COVID-19,
3. diagnosis of coma, vegetative state or minimally conscious state per Glasgow Coma Scale (GCS) at time of enrollment (excluding confounders such as sedation) and
4. clinical team plan for an MRI for clinical management.

Exclusion Criteria:

A subject with any of the following MRI contraindications will not be eligible for this study:

* electrical implants such as cardiac pacemakers or perfusion pumps
* ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
* ferromagnetic objects such as jewelry or metal clips in clothing that cannnot be easily removed for scanning
* pregnant volunteers

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Survivors of severe COVID-19 who have disorders of consciousness
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Disability Rating Scale score | 6 months
  Functional outcome measure. Maximum score of 29 represents high disability, minimum score of 0 represents no disability. Higher scores represent higher level of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fischer D, Threlkeld ZD, Bodien YG, Kirsch JE, Huang SY, Schaefer PW, Rapalino O, Hochberg LR, Rosen BR, Edlow BL. Intact Brain Network Function in an Unresponsive Patient with COVID-19. Ann Neurol. 2020 Oct;88(4):851-854. doi: 10.1002/ana.25838. Epub 2020 Aug 6. PMID 32613682
- [Derived] Fischer D, Snider SB, Barra ME, Sanders WR, Rapalino O, Schaefer P, Foulkes AS, Bodien YG, Edlow BL. Disorders of Consciousness Associated With COVID-19: A Prospective Multimodal Study of Recovery and Brain Connectivity. Neurology. 2022 Jan 18;98(3):e315-e325. doi: 10.1212/WNL.0000000000013067. Epub 2021 Dec 3. PMID 34862317